CLINICAL TRIAL: NCT00750425
Title: A Phase I, Open Label, Non-Randomised Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of Multiple Oral Doses of Cediranib (AZD2171, RECENTINÔ), in Patients With Advanced Solid Tumours
Brief Title: Phase 1 Study of the Effect of Ketoconazole on the PK of Multiple Doses of Cediranib in Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jane Robertson, Medical Science Director, RECENTIN, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8480C00020; EUDRACT number 2008-002271-27
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Advanced Solid Tumors
Keywords: advanced cancer,; metastatic; ketoconazole; pharmacokinetics; Phase I
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Cediranib alone, followed by cediranib plus ketoconazole, followed by cediranib alone
  Interventions: Drug: cediranib (RECENTIN TM, AZD2171)

INTERVENTIONS:
Drug: cediranib (RECENTIN TM, AZD2171) — 20 mg cediranib once daily from Days 1 to 7; then 20 mg cediranib plus 400 mg ketoconazole from Days 8-10; then 20 mg cediranib once daily from Days 11-23. At Day 24 patients may dose escalate to 30 mg tablet once daily providing the treatment is well tolerated (this may be escalated up to 45 mg if the 30mg dose is tolerated for a minimum of 14 days)

SUMMARY:
Phase I, open study to assess the effect of ketoconazole, a marketed drug, on the way the body handles the experimental drug cediranib, in patients with advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histological or cytological confirmation of advanced solid tumour (with the exception of prostate cancer), which is refractory to standard therapies or for which no standard therapy exists.
* Estimated life expectancy of at least 8 weeks
* WHO performance status (PS) 0-2.

Exclusion Criteria:

* Unstable brain/meningeal metastases
* Biochemistry/haematology results outside of required ranges
* History of significant GI impairment
* Inadequate bone marrow reserve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To assess the steady-state PK parameters of cediranib in the presence and absence of ketoconazole. | PK assessments to be taken until Day 42. Days 7 and 10 PK parameters used to assess the primary variables.

SECONDARY OUTCOMES:
Safety and tolerability of cediranib in the presence of ketoconazole by assessment of Adverse events (AEs) Laboratory findings,Vital signs, physical examination and Electrocardiogram. | Until study drug is discountinued

CONTACTS AND LOCATIONS:
Overall Officials: Jane Roberston, Study Director — AstraZeneca Aderley Park; Dr U Lassen, MD PhD, Principal Investigator — The Finsen Center, Copenhagen, Denmark
Locations (5):
- Canada (3):
  - Research Site, Hamilton
  - Research Site, Toronto
  - Research Site, Vancouver
- Denmark (2):
  - Research Site, Copenhagen
  - Research Site, Herlev